CLINICAL TRIAL: NCT00370734
Title: Effect of Percutaneous Botulinum Toxin A Injection on Natural Course of Upper Lid Retraction in Thyroid Eye Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8375
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Eye Diseases
Keywords: botulinum toxin; thyroid eye disease; lid retraction
MeSH Terms: conditions — Eye Diseases; Graves Ophthalmopathy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Botulinum toxin A injection

SUMMARY:
In active phase of thyroid eye disease some patients have obvious upper lid retraction , and sometimes exposure keratopathy .To date there is not any standard treatment for this situation . We are going to compare the natural course of the upper lid retraction with injection of botulinum toxin A injection to upper lid percutaneously.

ELIGIBILITY:
Inclusion Criteria:

* all the patients wiht oper lid retraction in active phase of thyroid ophthalmopathy

Exclusion Criteria:

* patients in non active phase

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2005-05; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Babak Babsharif, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Babak Babsharif, MD, Tehran, Tehran Province, Iran